CLINICAL TRIAL: NCT01562002
Title: Advanced Therapy for Ocular Surface Reconstruction. Allogenic Limbus Epithelial Stem-cell Transplant vs Bone Marrow Mesenchymal Stem-cell Transplant in Limbus Insufficiency Syndrome. Double-masked Randomized Trial
Brief Title: Safety Study of Stem Cell Transplant to Treat Limbus Insufficiency Syndrome
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA (Other)
Collaborators: University of Valladolid (Other); Centro en Red de Medicina Regenerativa de Castilla y Leon (Other); Red de Terapia Celular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IOBA-05-2010
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Limbus Corneae Insufficiency Syndrome
Keywords: limbus; cornea; insufficiency syndrome; stem cell transplant
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Bone Marrow mesenchymal stem cell (Experimental): Allogenic Bone Marrow mesenchymal stem cell in amniotic membrane transplant
  Interventions: Procedure: Stem Cell with Amniotic Membrane Transplant
- Allogenic limbal stem cell Transplant (Active Comparator): Stem Cell with Amniotic Membrane Transplant
  Interventions: Procedure: Stem Cell with Amniotic Membrane Transplant

INTERVENTIONS:
Procedure: Stem Cell with Amniotic Membrane Transplant — Single stem cell expansion in amniotic membrane transplant

SUMMARY:
The purpose of the study is to determine whether allogenic bone marrow stem cell transplant is safe and effective in the treatment of limbus insufficiency syndrome versus allogenic limbus stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female older than 18 years.
* Signed Informed consent
* Negative pregnancy test at inclusion for any potential childbearing female.
* Compromise of contraceptive method during all trial for any potential childbearing female.
* Diagnosis of Ocular Surface Failure due to Limbus Insufficiency Syndrome, based in any of the published characteristics as corneal surface neovascularization, loss of corneal transparency, epithelial irregularities, history of punctate keratitis, erosions or repetitive ulcers and presence of symptoms and confirmed by the presence of epithelial phenotype cells assessed with conjunctival impression cytology.
* Availability for all the scheduled visits during the study

Exclusion Criteria:

* Uncontrolled systemic disease (e.g. hypertension or diabetes) or any disease that under medical decision might put the patient at risk during the surgery or follow-up examinations or may cause any hazard in data analysis.
* Active ocular infection in any eye. If the infection can be cured, inclusion can be considered after 30 days of inactive infection since its end.
* Alterations in lid statics / dynamics or any other pathology (e.g. severe dry eye syndrome) except the one that originated the Limbus Insufficience that under medical opinion might alter the results. Any of these must be corrected 3 months prior to patient inclusion, before reconsidering rescreening.
* Limbus insufficiency syndrome which has not been previously treated with all medical (not surgical) procedures available.
* No availability for all scheduled visits during the study.
* Any other circumstance under investigator´s opinion that prevents patient inclusion even though normal inclusion and exclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Viability and safety of mesenchymal stem cell transplant | 1 Year
  Absence of cell metaplasia with phenotype different to corneal or conjunctival as expected, confirmed by corneal impression cytology and in vivo confocal laser ophthalmoscopy

SECONDARY OUTCOMES:
Absence of complications in pre and peri surgical implantation | 1 Week
  Correct handling and implantation of stem cell with amniotic membrane transplant following an 4 step classification.
Improvement of 2 lines in Best Corrected Visual Acuity | 12 month
  Improvement in visual acuity compared to baseline values before transplant

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Calonge, MD, PhD, Principal Investigator — Instituto Universitario de Oftalmobiología Aplicada (Institute of Applied Ophthalmobiology) - IOBA
Locations (1):
- IOBA, Valladolid, Valladolid, Spain

REFERENCES:
- [Derived] Perez I, Galindo S, Lopez-Miguel A, Nieto-Miguel T, de la Mata A, Lopez-Paniagua M, Alberca M, Herreras JM, Calonge M. In Vivo Confocal Microscopy in Limbal Stem Cell Deficiency After Mesenchymal Stem Cell Transplantation: A Sub-analysis from a Phase I-II Clinical Trial. Ophthalmol Ther. 2023 Dec;12(6):3251-3262. doi: 10.1007/s40123-023-00809-7. Epub 2023 Sep 29. PMID 37773479
- [Derived] Calonge M, Perez I, Galindo S, Nieto-Miguel T, Lopez-Paniagua M, Fernandez I, Alberca M, Garcia-Sancho J, Sanchez A, Herreras JM. A proof-of-concept clinical trial using mesenchymal stem cells for the treatment of corneal epithelial stem cell deficiency. Transl Res. 2019 Apr;206:18-40. doi: 10.1016/j.trsl.2018.11.003. Epub 2018 Nov 22. PMID 30578758